CLINICAL TRIAL: NCT02015637
Title: A Comparative Evaluation of the Single-dose Efficacy of Oral Delafloxacin Versus the Single-dose Efficacy of an Intramuscular Injection of Ceftriaxone in Subjects With Uncomplicated Urogenital Gonorrhea
Brief Title: Comparison of Delafloxacin Versus Ceftriaxone for the Treatment of Uncomplicated Gonorrhea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Melinta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML-3341-304
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-05

CONDITIONS: Gonorrhea
Keywords: Gonorrhea; N. gonorrhoeae; bacterial infection; Anti-Infective Agents; Anti-Bacterial Agents
MeSH Terms: conditions — Gonorrhea; Bacterial Infections | interventions — delafloxacin; Ceftriaxone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delafloxacin (Experimental): 900mg orally (2 x 450 mg tablets) administered once
  Interventions: Drug: Delafloxacin
- ceftriaxone (Active Comparator): Ceftriaxone 250 mg intramuscular injection administered once
  Interventions: Drug: Ceftriaxone

INTERVENTIONS:
Drug: Delafloxacin — single dose
  Arms: Delafloxacin
Drug: Ceftriaxone — single dose
  Arms: ceftriaxone

SUMMARY:
The purpose of this study is to evaluate the effects of a single oral dose of delafloxacin versus a single intramuscular injection of ceftriaxone in subjects with uncomplicated cervical, urethral, rectal, or pharyngeal gonorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female 15 years of age or older.
* Subject must have had 1 or more of the following occur:

  1. gonorrhea with the nucleic acid amplification test (NAAT) or culture within the previous 14 days
  2. unprotected genital contact within 14 days with a person confirmed to be infected with gonorrhea,
  3. gram-negative present in urogenital gram strain or male subject must present with purulent urethritis or a female subject with must present with mucopurulent cervical discharge
* Subject agrees to avoid unprotected sexual contact in order to minimize the risk of gonorrhea reinfection
* Subject must be in good health (ie, based on medical history), as determined by the investigator.
* In the opinion of the investigator, the subject must be able and willing to comply with protocol requirements. The subject must agree to provide reliable, verifiable contact information and agree to return for the Test-of-Cure Visit.
* If a subject's age is 15 years to less than the legal age of consent,a written, voluntarily signed assent must be obtained from the subject and a written, voluntarily signed informed consent must be signed by the subject's parent or legal guardian before the initiation of any study related procedures, unless the Institutional Review Board (IRB)/Independent Ethics Committee (IEC) determines that parent/legal guardian consent is not required.

Exclusion Criteria:

* Confirmed, or suspected, complicated or systemic gonococcal infection, such as pelvic inflammatory disease, arthritis, or endocarditis.
* Subject has taken one of the following products within 6 hours of the Entry Visit that may interfere with the absorption of a quinolone antibiotic: magnesium/aluminum antacids; sucralfate; Videx® (didanosine) chewable/buffered tablets; other highly buffered drugs; or other products containing calcium, iron, or zinc.
* Use of systemic or intravaginal antibiotics that are potentially effective against gonorrhea 4 weeks prior to study drug administration.
* Subjects with a current or prior history of seizures, and subjects being treated with drugs that are known to have a sizable potential of or reduce the threshold for inducing seizures (eg, bupropion, theophylline, and tricyclic and tetracyclic antidepressants).
* Current use of systemic corticosteroid or immunosuppressive drugs.
* Known significant immunosuppression (eg, cluster of differentiation (CD4) cell count <200/mm3 or absolute neutrophil count <500/mL).
* Cytotoxic chemotherapy or radiation therapy during the previous 3 months.
* Subject is co-infected with an additional sexually transmitted disease (STD) for which treatment cannot be safely deferred until after the Test-of-Cure Visit unless the treatment is not potentially effective against gonorrhea.
* Subject has used an investigational drug or product within 30 days before study drug dosing.
* Medical history of Type 1 hypersensitivity to antibiotics of the quinolone or cephalosporin classes.
* Hysterectomized subjects without a cervix are ineligible.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sue Cammarata, MD, Study Director — Melinta Therapeutics, Inc.
Locations (25):
- United States (25):
  - Melinta 304 Study, Birmingham, Alabama
  - Melinta 304 Study Site, Chula Vista, California
  - Melinta 304 Study Site, La Mesa, California
  - Melinta 304 Study Site, Los Angeles, California
  - Melinta 304 Study Site, San Francisco, California
  - Melinta 304 Study, Atlanta, Georgia
  - Melinta 304 Study, Decatur, Georgia
  - Melinta 304 Study Site, Indianapolis, Indiana
  - Melinta 304 Study Site, New Orleans, Louisiana
  - Melinta 304 Study Site, Omaha, Nebraska
  - Melinta 304 Study Site, Las Vegas, Nevada
  - Melinta 304 Study Site, Brooklyn, New York
  - Melinta 304 Study, Brooklyn, New York
  - Melinta 304 Study Site, New York, New York
  - Melinta 304 Study Site, The Bronx, New York
  - Melinta 304 Study Site, Durham, North Carolina
  - Melinta 304 Study Site, Greensboro, North Carolina
  - Melinta 304 Study Site, Cleveland, Ohio
  - Melinta 304 Study Site, Columbus, Ohio
  - Melinta 304 Study Site, Portland, Oregon
  - Melinta 304 Study, Erie, Pennsylvania
  - Melinta 304 Study Site, Philadelphia, Pennsylvania
  - Melinta 304 Study Site, Pittsburgh, Pennsylvania
  - Melinta 304 Study Site, Houston, Texas
  - Melinta 304 Study Site, Seattle, Washington

REFERENCES:
- [Derived] Hook EW 3rd, Golden MR, Taylor SN, Henry E, Tseng C, Workowski KA, Swerdlow J, Nenninger A, Cammarata S. Efficacy and Safety of Single-Dose Oral Delafloxacin Compared With Intramuscular Ceftriaxone for Uncomplicated Gonorrhea Treatment: An Open-Label, Noninferiority, Phase 3, Multicenter, Randomized Study. Sex Transm Dis. 2019 May;46(5):279-286. doi: 10.1097/OLQ.0000000000000971. PMID 30985632

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Delafloxacin | Ceftriaxone
Started | 306 | 154
Completed | 298 | 149
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 3 | 5
Not completed — Adverse Event | 3 | 0
Not completed — Did not take study drug | 2 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Delafloxacin | Ceftriaxone | Total
Number analyzed (Participants) | 304 | 154 | 458
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (8.82) | 28.7 (10.04) | 29.3 (9.25)
Age, Customized [Count of Participants; unit: Participants]
  <18 year | 1 | 2 | 3
  18-70 years | 303 | 152 | 455
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: This information was collected on males only.
  Participants
    Men who:: number analyzed (Participants) | 245 | 119 | 364
    Men who:: Were heterosexul | 132 | 59 | 191
    Men who:: Had sex with men or were bisexual | 112 | 60 | 172
    Men who:: Missing | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 35 | 94
  Male | 245 | 119 | 364
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 22 | 56
  Not Hispanic or Latino | 268 | 131 | 399
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 186 | 92 | 278
  White | 98 | 48 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 13 | 25
Positive culture for Gonorrhea (GC) [Count of Participants; unit: Participants] — Positive culture for N gonorrhoeae obtained from 1 or more anatomical sites (i.e., urogenital, pharyngeal, rectal) at the Entry Visit, i.e. were part of the Microbiological Intent-to-treat (MITT) population.
  Participants | 239 | 107 | 346

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Cure or Failure of Urogenital Gonorrhea at Test of Cure (TOC) in the Urogenital MITT (UMITT) Population
Description: Cure for the primary outcome measure was defined as the eradication of N. gonorrhoeae at TOC as determined by a negative culture obtained from the urogenital site, which was positive at study entry, and with no additional antibiotics with activity against N. gonorrhoeae being administered from study entry through TOC.
Time Frame: Day 7 (± 3 days)
Population: The primary efficacy analysis was done on the UMITT population, which included all subjects in the ITT analysis set who had a positive culture for N gonorrhoeae obtained at a urogenital site at the Entry Visit, and who did not receive antibiotic therapy for a C trachomatis infection that was potentially effective against N gonorrhoeae prior to TOC.
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Ceftriaxone
Number analyzed (Participants) | 228 | 100
Participants
  Cure | 194 | 91
  Failure | 34 | 9
Statistical Analysis 1: Comparison: Delafloxacin vs Ceftriaxone; Test type: Non-Inferiority — Two-sided 95% confidence intervals (CIs) using the Wald test was constructed for comparisons between delafloxacin and ceftriaxone. A hierarchical approach was implemented for the primary and secondary analyses to control for the overall type 1 error rate of 0.05 due to multiple comparisons; Difference in cure rate = -5.9, 95% CI 2-sided [-13.18 to 1.36]

2. Secondary Outcome: Number of Subjects With Cure or Failure of Urogenital Gonorrhea at Test of Cure (TOC) in the Urogenital Microbiologically Evaluable (UME) Population
Description: Cure for the seconday outcome measure was defined as the eradication of N. gonorrhoeae at TOC as determined by a negative culture obtained from the urogenital site, which was positive at study entry, and with no additional antibiotics with activity against N. gonorrhoeae being administered from study entry through TOC.
Time Frame: Day 7 (± 3 days)
Population: Urogenital ME (UME): All subjects included in the UMITT analysis set who received study drug and had no important protocol deviations that would affect the assessment of efficacy
Measure: Count of Participants; unit: Participants
Arm/Group | Delafloxacin | Ceftriaxone
Number analyzed (Participants) | 226 | 95
Participants
  Cure | 194 | 91
  Failure | 32 | 4
Statistical Analysis 1: Comparison: Delafloxacin vs Ceftriaxone; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Difference in cure rates = -9.9, 95% CI 2-sided [-16.03 to -3.87]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring from the time the subject signed the Informed Consent Form (ICF) through the follow-up phone contact were reported and followed to resolution. Collection of all AEs occurred from the time the subject received study drug (Day 1) through the TOC visit (Day 7 +/- 3), or up to 10 days. Only Serious Adverse Events (SAEs) were collected after the TOC visit through the follow-up phone contact (Day 30 +/- 3 days), or up to 33 days.
Description: AEs were reported in the Safety Population which was defined as all subjects that received study drug. Two patients that were in the ITT population (all subjects randomly assigned to a treatment group) for delafloxacin did not receive study drug.
Arm/Group | Delafloxacin | Ceftriaxone
All-Cause Mortality (participants affected / at risk) | 0/304 | 0/154
Serious Adverse Events (participants affected / at risk) | 0/304 | 1/154
Other Adverse Events (participants affected / at risk) | 121/304 | 13/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delafloxacin (N=304) | Ceftriaxone (N=154)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Delafloxacin (N=304) | Ceftriaxone (N=154)
Diarrhea (Gastrointestinal disorders) | 97 | 11
Nausea (Gastrointestinal disorders) | 24 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Melinta has the right to first publication of results, which would be made in conjunction with the PIs from all appropriate sites. Thereafter, PIs may publish results provided the PI submits the proposed publication to Melinta for review at least 60 days prior to the date of the proposed publication. Melinta may remove any information that is considered confidential and/or proprietary. If a publication is not submitted within 12 months of study conclusion, the PI may publish results.